CLINICAL TRIAL: NCT05054465
Title: A Phase 1b-2 Trial to Assess the Safety and Efficacy of a Venetoclax and Navitoclax Consolidation in High-risk Patients With T- Cell Acute Lymphoblastic Leukemia Prior to Allogeneic Transplantation Followed by Venetoclax and Navitoclax Post-transplant Maintenance
Brief Title: A Phase 1b-2 Trial to Assess Venetoclax and Navitoclax Consolidation and Post-transplant Maintenance in High-risk Patients With T-ALL
Acronym: ITALLI001
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Israeli Medical Association (Other)
Collaborators: Rabin Medical Center (Other); Sheba Medical Center (Other Government); Rambam Health Care Campus (Other); Tel Aviv Medical Center (Other); Soroka University Medical Center (Other); Shaare Zedek Medical Center (Other); Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITALLI001
Record Dates: First submitted 2021-06-10; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-06

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — navitoclax; venetoclax

STUDY DESIGN:
Intervention Model Description: A national, multicenter, phase II clinical trial to evaluate the benefit of pre-transplant (alloSCT) consolidation (cons.) and post-alloSCT maintenance with navitoclax (NAV) and venetoclax (VEN) in patients with T-ALL, LBL and MPAL T/M in CR1 designated for alloSCT. Pre-alloSCT cons. with VEN and NAV: Patients will be treated with VEN 400 mg QD and NAV 50mg QD according to the RP2D presented by Pullarkat et al. (doi: 10.1158/2159-8290.CD-20-1465) for two 28 day cycles. Following 2 cycles re-staging marrow including MRD assessment and imaging will be followed by alloSCT according to local protocol. Post-alloSCT maintenance with VEN and NAV: Within 90 days from alloSCT patients will be started on VEN and NAV maintenance. For post-alloSCT maintenance a dose escalation scheme based on the BOIN design will be applied with a maximal dose of VEN 400 mg QD and NAV 50mg QD according to the RP2D presented by Pullarkat et al.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pre-transplant consolidation and post-transplant maintnance with navitoclax and venetoclax. (Experimental): Patients will be treated with VEN 400 mg QD and NAV 50mg QD according to the RP2D presented by Pullarkat et al. (doi: 10.1158/2159-8290.CD-20-1465) for two 28 day cycles. Following 2 cycles re-staging marrow including MRD assessment and imaging will be followed by alloSCT according to local protocol.Within 90 days from alloSCT patients will be started on VEN and NAV maintenance. For post-alloSCT maintenance a dose escalation scheme based on the BOIN design will be applied with a maximal dose of VEN 400 mg QD and NAV 50mg QD according to the RP2D presented by Pullarkat et al.
  Interventions: Drug: Navitoclax; Drug: Venetoclax

INTERVENTIONS:
Drug: Navitoclax — P.O 50mg QD Q28 days for 2 cycles pre-transplant Up to 50mg QD Q28 days maintnance post-transplant based on MTD
Drug: Venetoclax — P.O 400mg QD Q28 days for 2 cycles pre-transplant Up to 400mg QD Q28 days maintnance post-transplant based on MTD

SUMMARY:
This is a national, multicenter, phase II clinical trial to evaluate the potential benefit of pre-transplant consolidation and post-transplant maintenance with navitoclax and venetoclax in patients with T-ALL, LBL and MPAL T/M in first complete remission designated for allogeneic transplantation.

Pre-transplantation consolidation with venetoclax and navitoclax:

Patients in CR designated for transplantation will be treated with venetoclax 400 mg QD and navitoclax 50mg QD according to the RP2D presented by Pullarkat et al. (Cancer Discov . 2021 Feb 16;candisc.1465.2020. doi: 10.1158/2159-8290.CD-20-1465.) for two 28 day cycles. Following 2 cycles re-staging marrow including MRD assessment and imaging as need will be followed by alloSCT according to local protocol.

Post-transplantation maintenance with venetoclax and navitoclax:

Within 90 days from alloSCT patients will be started on venetoclax and navitoclax maintenance.

Due to lack of data regarding the toxicity of navitoclax and venetoclax in the ALL post alloSCT maintenance setting a dose escalation scheme based on the BOIN design will be applied as outlined (TBD) with a maximal dose of venetoclax 400 mg QD and navitoclax 50mg QD according to the RP2D presented by Pullarkat et al. (Cancer Discov . 2021 Feb 16;candisc.1465.2020. doi: 10.1158/2159-8290.CD-20-1465).

DETAILED DESCRIPTION:
Despite several therapeutic advancements, the outcome of adults with T-cell acute lymphoblastic leukemia (ALL) and lymphoblastic lymphoma (LBL) remains unsatisfactory, especially in those patients with high-risk disease features.

In such high-risk patients, allogenic transplantation is usually recommended, when feasible. Interventions to increase response and survival are needed for this high-risk subset of patients.

In pre-clinical studies, certain T-cell ALL cell lines were shown to be particularly sensitive to BCL2 inhibition (Peirs et al, Blood 2014). Recent reports demonstrate that venetoclax in combination with navitoclax is an effective approach to patients with relapsed/refractory ALL (Lacayo. ASH 2019. Abstr 285). Venetoclax in combination with chemotherapy in elderly patients with ALL also demonstrated promising efficacy with preliminary reasonable safety signals (Jain. ASH 2019. Abstr 3867). We hypothesize that adding venetoclax and navitoclax as a pre-transplant intervention and as maintenance may improve post-transplant outcome for these patients.

The primary objectives of this study are:

1. To evaluate the efficacy of venetoclax in combination with navitoclax consolidation in newly diagnosed T-ALL patients prior to alloSCT.
2. To evaluate the safety and potential benefit of post-transplant venetoclax and navitoclax maintenance therapy in patients with T-ALL.

The secondary objectives of this study are:

1. To evaluate the impact of pre-transplant venetoclax/navitoclax consolidation.

This is a national, multicenter, phase II clinical trial to evaluate the potential benefit of pre-transplant consolidation and post-transplant maintenance with navitoclax and venetoclax in patients with T-ALL, LBL and MPAL T/M in first complete remission designated for allogeneic transplantation.

Pre-transplantation consolidation with venetoclax and navitoclax:

Patients in CR designated for transplantation will be treated with venetoclax 400 mg QD and navitoclax 50mg QD according to the RP2D presented by Jabbour et al. (EHA25; S116) for two 28 day cycles. Following 2 cycles re-staging marrow including MRD assessment and imaging as need will be followed by alloSCT according to local protocol.

Post-transplantation maintenance with venetoclax and navitoclax:

Within 90 days from alloSCT patients will be started on venetoclax and navitoclax maintenance.

Due to lack of data regarding the toxicity of navitoclax and venetoclax in the ALL post alloSCT maintenance setting a dose escalation scheme based on the BOIN design will be applied as outlined (TBD) with a maximal dose of venetoclax 400 mg QD and navitoclax 50mg QD according to the RP2D presented by Jabbour et al. (EHA25; S116).

The BOIN design will be based on the cumulative number of subjects who experience a dose-limiting toxicity (DLT) at a particular dose level. Dose escalation decisions will be based on 3-6 DLT-evaluable subjects at each dose level. At least 6 subjects will be treated during dose escalation and assessed for safety at what is ultimately used for expansion.

Planned follow up is durring maintnance every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the informed consent document.
2. Have a documented new diagnosis of T-ALL, T-LBL or MPAL T/Myeloid according to the WHO 2016 classification.
3. Patients in first complete response that are planned for an alloSCT.
4. Patient induction with a BFM backbone, asparginase containing induction.
5. Adequate bone marrow reserve; • Absence of growth factors, thrombopoietic factors, or platelet transfusions in the week prior to day 1 of therapy with Navitoclax and venetoclax.

   * Platelet count ≥ 50 × 109 /L
   * Absolute neutrophil count (ANC) ≥ 1 × 109 /L.
6. Hepatic function and enzymes:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 × ULN (exception: subjects with Gilbert's Syndrome may have total bilirubin > 1.5 × ULN)
   * Coagulation: activated partial thromboplastin time (aPTT) and international normalized ratio (INR) ≤ 1.5 × ULN.
7. Renal function: calculated creatinine clearance ≥ 30 mL/min

• For the post-transplant maintenance phase:Patient should satisfy all the above criteria.

• Patient must not have grade 2 or higher for aGvHD and moderate or severe for cGvHD.

9. Females of childbearing potential (FCBP) may participate, providing they meet the following conditions: Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study, and for 3 months following EOT; and have a negative serum or urine pregnancy test (investigator's discretion; sensitivity at least 25 mIU/mL) at screening; and have a negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting study therapy in the treatment phase (note that the screening serum pregnancy test can be used as the test prior to starting study therapy in treatment phase if it is performed within the 72-hour timeframe).

10. Male subjects with a female partner of childbearing potential must agree to the use of at least two physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study and for 3 months following the last dose of study drug.

11. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

12. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Age <18 at the time of signing the informed consent document.
2. Ph-positive disease.
3. Patient not regarded as candidates for allogeneic transplantation.
4. Non-BFM based, asparginase containing induction (including HyperCVAD)
5. Concomitant Medications:

   * Subject must not have been treated with a medical product without any global regulatory approvals within 30 days or 5 half-lives of the drug (whichever is shorter) prior to Cycle 1 Day 1 and must not be currently receiving AML treatment in another clinical interventional study.
   * Cytochrome P450 (CYP)3A inducers and grapefruit/grapefruit products: Subject must not have received a known strong or moderate CYP3A inducer 7 days prior to Cycle 1 Day 1. Subject must not have known medical conditions requiring chronic therapy of moderate CYP3A inducers.
   * Cytochrome P450 (CYP)3A inhibitors: Subject must not have received a known strong or moderate CYP3A inhibitors 7 days prior to Cycle 1 Day 1. Subject must not have known medical conditions requiring chronic therapy of strong or moderate CYP3A inhibitors (appendix 2).
   * Subject must not have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or starfruit within 3 days prior to Cycle 1 Day 1.
   * Subject must not have received any live vaccine within 4 weeks prior to Cycle 1 Day 1.
   * The subject must not be expected to need a live vaccination throughout study participation.
   * The subject must not be expected to need a live vaccine in case of the following 7 conditions:

1. Less than 24 months following transplantation 2. Active GvHD 3. Lymphocyte count < 1,500/μL 4. Less than 12 months in remission 5. Less than 3 months after the last dose of oncological therapy 6. Less than 4 weeks after the most recent infusion of immunoglobulins 7. Less than 4 weeks after the most recent immunosuppressive therapy

• Subject must not have been treated with any investigational drug within 30 days prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study

6. Known Human Immunodeficiency Virus (HIV).

7. No history of being positive for hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Inactive hepatitis carrier status or low viral hepatitis titers on antivirals (non-exclusionary medications) are not excluded.

8. Known or suspected hypersensitivity to any of the study drugs.

9. Pregnant or lactating females.

10. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.

11. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.

12. Participation to an investigational drug trial in the last month before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  EFS is defined for all patients and measured from the date of entry on study. It is measured until treatment failure defined as molecular or morphological relapse from CR, treatment discontinuation due to drug related toxicity or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
Frequency of AE's during therapy | Recorded every 3 months for 2 years during follow up
  AE's based on CTCAE 5.0
Rate of grade 3-4 GvHD events | 90 days
  GvHD rate at 90 days - defined as Grade 3 or higher for aGvHD and moderate or severe for cGvHD as defined by the investigator following National Institutes of Health (NIH) criteria.
Minimal Residual Disaease status | Recorded every 3 months for 2 years during follow up
  Frequency of MRD negativity at the following time points: post induction II (week 12), after cycle 1 of-venetoclax and navitoclax therapy, after cycle 2 and before alloSCT and Q3 months post transplant (centrally assessed by PCR)

CONTACTS AND LOCATIONS:
Locations (6):
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pullarkat VA, Lacayo NJ, Jabbour E, Rubnitz JE, Bajel A, Laetsch TW, Leonard J, Colace SI, Khaw SL, Fleming SA, Mattison RJ, Norris R, Opferman JT, Roberts KG, Zhao Y, Qu C, Badawi M, Schmidt M, Tong B, Pesko JC, Sun Y, Ross JA, Vishwamitra D, Rosenwinkel L, Kim SY, Jacobson A, Mullighan CG, Alexander TB, Stock W. Venetoclax and Navitoclax in Combination with Chemotherapy in Patients with Relapsed or Refractory Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma. Cancer Discov. 2021 Jun;11(6):1440-1453. doi: 10.1158/2159-8290.CD-20-1465. Epub 2021 Feb 16. PMID 33593877